CLINICAL TRIAL: NCT00698087
Title: Study to Compare the Safety, Immunogenicity and Reactogenicity of Different Formulations of GSK Biologicals' (Previously SmithKline Beecham Biologicals') MPL-Adjuvanted Recombinant Hepatitis B Vaccine to That of Engerix™-B
Brief Title: Comparison of Safety, Immuno- and Reactogenicity of MPL-Adjuvanted Recombinant Hepatitis B Vaccine to That of Engerix™-B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Isabelle Harpigny, GSK
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 208129/016
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Last update posted 2008-06-16 (Estimated); Status verified 2008-06

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Engerix™-B; Adjuvanted recombinant hepatitis B vaccine
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Group A (Experimental)
  Interventions: Biological: MPL-Adjuvanted recombinant hepatitis B vaccine
- Group B (Active Comparator)
  Interventions: Biological: Engerix™-B
- Group C (Experimental)
  Interventions: Biological: MPL-Adjuvanted recombinant hepatitis B vaccine

INTERVENTIONS:
Biological: MPL-Adjuvanted recombinant hepatitis B vaccine — Intramuscular injection, 2 or 3 doses, 2 different formulations
  Arms: Group A; Group C
Biological: Engerix™-B — Intramuscular injection, 2 or 3 doses
  Arms: Group B

SUMMARY:
The purpose of the study is to compare the safety, reactogenicity and immunogenicity of different formulations of adjuvanted recombinant hepatitis B vaccine to that of Engerix™-B when administered at 0, 2 months with a booster at month 12 if necessary

DETAILED DESCRIPTION:
At the time of conduct of this study, the sponsor GlaxoSmithKline was known by its former name SmithKline Beecham

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 40 years old.
* Written informed consent will have been obtained from the subjects.
* Good physical condition as established by physical examination and history taking at the time of entry.
* Female participants will avoid becoming pregnant during the study period and they will have been on a contraceptive program for at least 2 months before entry

Exclusion Criteria:

* Pregnancy or lactation.
* Positive titres for anti hepatitis B antibodies
* Any vaccination against hepatitis B in the past.
* Any previous administration of MPL.
* Elevated serum liver enzymes.
* History of significant and persisting hematologic, hepatic, renal, cardiac or respiratory disease.
* Axillary temperature > 37.5°C at the time of injection.
* Any acute disease at the moment of entry.
* Chronic alcohol consumption.
* Any treatment with immunosuppressive or immunostimulant therapy.
* Any chronic drug treatment, which in the investigator's opinion, precludes inclusion into the study.
* History of allergic disease likely to be stimulated by any component of the vaccine.
* Simultaneous administration of any other vaccine(s).
* Administration of any immunoglobulin during the study period.
* Simultaneous participation in any other clinical trial

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 1995-01; Primary Completion 1996-02 (Actual); Study Completion 1996-02 (Actual)

PRIMARY OUTCOMES:
Anti-HBs antibody concentrations | At M3 and M13
Occurrence of local and general solicited symptoms | 4-day follow-up after vaccination
Occurrence of unsolicited symptoms | 30-day follow-up after vaccination

SECONDARY OUTCOMES:
SAEs | Throughout the study up to 30 days after last vaccination
Anti-HBs antibody concentrations | Months 2, 3, 6, 9, 12, 13

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Clinical Trials Call Center, Vienna, Austria